CLINICAL TRIAL: NCT04978155
Title: Usefulness of Doppler Ultrasound Carried Out by the Vascular Surgeon After Loco-regional Anesthesia for Preferred Access
Status: Completed | Type: Observational
Sponsor: University Paul Sabatier of Toulouse (Other)
Responsible Party: Principal Investigator, Aurélien Hostalrich, Vascular Surgeon,MD, Principal investigator, University Paul Sabatier of Toulouse
Other Study IDs: ECHO FAV
Record Dates: First submitted 2021-07-09; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Arterio-venous Fistula
Keywords: Arterio-veinous fistula access; preoperative Doppler ultrasound; maturation access
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Echo group: All the patients (n=90) who had an AVF creation with preoperative venous identification by the surgeon at CHU de TOULOUSE (echo group).
  Interventions: Diagnostic Test: Duplex ultrasound performed by the surgeon after locoregional anesthesia
- Control: All the patients (n=93) who had a native AVF placed during the year 2019 without having received immediate preoperative ultrasound and therefore there was no alteration in the surgical project in relation to that planned at the time of the consultation

INTERVENTIONS:
Diagnostic Test: Duplex ultrasound performed by the surgeon after locoregional anesthesia — Just after locoregional anesthesia, the surgeon perform a duplex ultrasound to determinate if the target vessel chosen to create the arterio-venous fistulae match with the pre-operative duplex performed during the consultation. So the plan can be changed such as more distal, more proximal creation, changing vein or artery target.
  Groups: Echo group

SUMMARY:
Preoperative vascular mapping with echo-Doppler is acknowledged as indispensable to create an arteriovenous fistula for haemodialysis (AVF). The conditions for performing this examination are not always ideal (venous vasospasm in cool temperatures, variability of the volume status in the dialysis patient).

On the other hand, the use of a loco-regional anaesthesia (LRA) results in the vasodilation of the limb thus rendering it possible to use the veins which were initially considered too small.

The aim of this study is to assess the functionality of our AVF when ultrasound identification was used by the surgeon after the LRA. These results have been compared with those of the preceding year during which this identification was not implemented.

DETAILED DESCRIPTION:
The investigators conducted a prospective study in the year 2020 during which all the patients (n=90) had an AVF creation with preoperative venous identification by the surgeon at university hospital of TOULOUSE (France)(echo group).

All the patients gave their consent, and the database was anonymised upon completion.

All patients were seen in a preoperative consultation with venous mapping carried out by a physician specialised in the use of Doppler ultrasonography. Following this consultation, a type of fistula was programmed in accordance with the Silva criteria (notably a vein with a diameter of over 2.5mm and an artery of 2mm). On the day of the operation, loco-regional anaesthesia was performed under sonographic guidance according to the previous description . The decision of the block approach and the choice of local aesthetic agent was left to the discretion of the anaesthesiologist.

The surgeon carried out an ultrasound and modification of the type of AVF was then made if the Silva criteria differed from those described during initial consultation. The modification could be a more distal creation, a more proximal creation, a change of vein or a change of artery.

The investigators succeeded to create more distal AVF when the vein had a diameter of over 2.5mm after LRA. Furthermore, the investigators reassembled the AVF when the vein appeared too small or residual (for example, following the attachment of an infusion having occurred between mapping and the surgery).

The same team of 4 surgeons participated in the creation of the AVF for both the echo group and the control group.

All patients were given a preoperative assessment of their heart function and cardiovascular risk factors (HTA, diabetes, smoking, dyslipidaemia). Prior strokes and coronary diseases were also registered as well as the patients' BMI and American society of anesthesiology score.

The definition of the good development of the haemodialysis access is based on the National Kidney Foundation's criteria: Blood flow>600ml, diameter over 6mm and lower depth of 6mm. On the other hand, permeability was based on the criteria of the Society for Vascular Surgery : primary permeability lasts from the creation to the first dilation episode or transposition of anastomosis required to maintain the access. Assisted primary permeability ends at the time of the first occlusion episode. Secondary permeability ends with the abandonment or the definitive withdrawal of the AVF due to failure.

The first postoperative consultation took place at around the 6th week after the creation which is the normal time necessary for the smooth development of an AVF .

The investigators compared all these results with our control group which consists of all the patients who had a native AVF placed during the year 2019 without having received immediate preoperative ultrasound and therefore there was no alteration in the surgical project in relation to that planned at the time of the consultation. Demographic data was similarly compiled and all the evaluation criteria compared

ELIGIBILITY:
Inclusion Criteria:

* Native AVF access
* During the year 2020
* Preoperative mapping during the consultation
* Loco-regional anesthesia

Exclusion Criteria:

* Redo surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients who had an AVF creation with preoperative venous identification by the surgeon at CHU de TOULOUSE during the year 2020.
Sampling Method: Non-Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Functionality of the AVF at the time of the postoperative | 6 weeks
  An AVF is defined as functional if all the criteria of the good development of the haemodialysis access (based on the National Kidney Foundation's criteria) are present : Blood flow>600ml, diameter over 6mm and lower depth of 6mm

SECONDARY OUTCOMES:
The rate of planning change between the surgical project at the time of the consultation and the AVF that is finally placed | During the surgery
Primary, assisted primary and secondary permeability of our accesses | 12 months
  permeability was based on the criteria of the Society for Vascular Surgery : primary permeability lasts from the creation to the first dilation episode or transposition of anastomosis required to maintain the access. Assisted primary permeability ends at the time of the first occlusion episode. Secondary permeability ends with the abandonment or the definitive withdrawal of the AVF due to failure

CONTACTS AND LOCATIONS:
Locations (1):
- aurelien Hostalrich, Toulouse, France

REFERENCES:
- [Derived] Hostalrich A, Boisroux T, Segal J, Lebas B, Ricco JB, Chaufour X. Assessment of Duplex Ultrasound Carried Out by the Vascular Surgeon After Locoregional Anesthesia for Preferred Arteriovenous Fistula Access. Ann Vasc Surg. 2022 Jul;83:117-123. doi: 10.1016/j.avsg.2021.11.014. Epub 2021 Dec 20. PMID 34942337